CLINICAL TRIAL: NCT02017405
Title: A Randomized, Crossover Clinical Study Evaluating the Digestibility of Serum-Derived Bovine Immunoglobulin Protein Isolate (SBI) in Healthy Adults
Brief Title: Study Evaluating the Digestibility of Serum-Derived Bovine Immunoglobulin Protein Isolate in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entera Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EH4001
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Digestibility; Healthy volunteers; serum-derived bovine immunoglobulin protein isolate; bovine IgG; adults

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5g Serum-derived bovine immunoglobulin protein isolate (SBI) (Other): Phase 1: Twelve subjects will receive either a 5.0 g total daily dose of SBI on Day 1 followed by 5.0 g Placebo on Day 2 or a 5.0 g total daily dose of Placebo on Day 1 followed by 5.0 g SBI on Day 2 during the double-blind, crossover phase.
  Phase 2: 2.5g SBI will be taken two times a day for 14 days during the open-label phase.
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
- 10g Serum-derived bovine immunoglobulin protein isolate (SBI) (Other): Phase 1: Twelve subjects will receive either a 10.0 g total daily dose of SBI on Day 1 followed by 10.0 g Placebo on Day 2 or a 10.0 g total daily dose of Placebo on Day 1 followed by 10.0 g SBI on Day 2 during the double-blind, crossover phase.
  Phase 2: 5.0 g SBI will taken two times a day for 14 days during the open-label phase.
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
- 20g Serum-derived bovine immunoglobulin protein isolate (SBI) (Other): Phase 1: Twelve subjects will receive either a 20.0 g total daily dose of SBI on Day 1 followed by 20.0 g Placebo on Day 2 or a 20.0 g total daily dose of Placebo on Day 1 followed by 20.0 g SBI on Day 2 during the double-blind, crossover phase.
  Phase 2: 20.0 g SBI will be taken two times a day for 14 days during the open-label phase.
  Interventions: Other: Serum-derived bovine immunoglobulin protein isolate (SBI)
- Matching Placebo (Other): Placebo will be taken either on Day 1 or on Day 2 based on the randomization during the double-blind, crossover phase.
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Other: Serum-derived bovine immunoglobulin protein isolate (SBI) — Serum-derived bovine immunoglobulin protein isolate is a specially formulated light-colored protein powder composed of immunoglobulin (IgG) and other serum proteins similar to those found in colostrum and milk. Serum-derived bovine immunoglobulin protein isolate does not contain any milk products such as lactose, casein, or whey. Serum-derived bovine immunoglobulin protein isolate is gluten-free, dye-free, and soy-free. Serum-derived bovine immunoglobulin protein isolate is manufactured in accordance with current Good Manufacturing Practice (cGMP) and FDA guidelines for medical food ingredients.
  Other Names: EnteraGam™
  Arms: 10g Serum-derived bovine immunoglobulin protein isolate (SBI); 20g Serum-derived bovine immunoglobulin protein isolate (SBI); 5g Serum-derived bovine immunoglobulin protein isolate (SBI)
Other: Matching Placebo
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to determine the digestibility of serum-derived bovine immunoglobulin protein isolate in healthy adults. The information generated may help elucidate SBI's mechanism of action.

DETAILED DESCRIPTION:
This study is evaluating the safety and absorption of serum-derived bovine immunoglobulin protein isolate (SBI) in healthy adults using 5, 10, and 20 g doses of SBI and placebo equivalents in a double blind crossover study and SBI affects over 14 days. Additionally, plasma amino acid response and IgG concentrations in both stool and plasma will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18-32
* Medically normal with no significant abnormal findings at screening

Exclusion Criteria:

* Allergy or intolerance to beef
* Participated in another investigational study within 30 days
* Seropostive for HIV, hepatitis B surface antigen, hepatitis C virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Weaver, PHD, Study Director — Entera Health
Locations (2):
- United States (2):
  - PMG Research of Cary, Cary, North Carolina
  - Wake Research Associates, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EnteraGam™ — http://www.enteragam.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1A: Crossover Phase:
  5.0g total daily dose of SBI on Day 1 followed by 5.0g Placebo on Day 2
  Open Label Phase:
  5.0g total daily dose of SBI will be taken for 14 days
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1B: Crossover Phase:
  5.0g total daily dose of Placebo on Day 1 followed by 5.0g SBI on Day 2
  Open Label Phase:
  5.0g total daily dose of SBI will be taken for 14 days
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2A: Crossover Phase:
  10.0g total daily dose of SBI on Day 1 followed by 10.0g Placebo on Day 2
  Open Label Phase:
  10.0g total daily dose of SBI will be taken for 14 days
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2B: Crossover Phase:
  10.0g total daily dose of Placebo on Day 1 followed by 10.0g SBI on Day 2.
  Open Label Phase:
  10.0g total daily dose of SBI will be taken for 14 days
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3A: Crossover Phase:
  20.0g total daily dose of SBI on Day 1 followed by 20.0g placebo on day 2.
  Open Label Phase:
  20.0g total daily dose of SBI will be taken for 14 days
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3B: Crossover Phase:
  20.0g total daily dose of Placebo on Day 1 followed by 20.0g SBI on Day 2
  Open Label Phase:
  20.0g total daily dose of SBI will be taken for 14 days
Period: Two-day, Double-blind, Crossover Phase
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1A | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1B | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2A | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2B | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3A | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3B
Started (Dosing errors occurred in six subjects during the double-blind, crossover phase. Four subjects assigned to 10g of SBI received 5g of SBI and two subjects assigned to 20g of SBI received 10g of SBI. An additional six subjects were added to the 2-day, double-blind, crossover phase to ensure ~12 subjects per SBI gram dosage group.) | 9 | 9 | 7 | 5 | 5 | 7
Completed | 9 | 9 | 7 | 5 | 5 | 6 (Patient withdrew after receiving placebo dose and prior to receiving 20g SBI dose.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Open-label Phase
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1A | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 1B | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2A | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 2B | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3A | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - 3B
Started (Dosing errors occurred in six subjects during the double-blind, crossover phase. These six subjects continued with the originally assigned dose of SBI for the 14-day, open-label phase of the study. This led to a difference in number of participants who completed phase 1 and started phase 2.) | 7 (No placebo in the open label phase) | 7 (No placebo in the open label phase) | 7 (No placebo in the open label phase) | 7 (No placebo in the open label phase) | 7 (No placebo in the open label phase) | 6 (No placebo in the open label phase)
Completed | 6 | 6 | 7 | 7 | 7 | 6
Not Completed | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | Total
Number analyzed (Participants) | 18 | 12 | 12 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (9.66) | 45.0 (16.64) | 39.9 (13.26) | 40.2 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 7 | 23
  Male | 8 | 6 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 17 | 12 | 12 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 3 | 2 | 15
  White | 7 | 9 | 9 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Total Plasma Amino Acids
Description: Plasma amino acid concentrations (umol/mL) were measured after administration of SBI or Placebo during the Cross-over phase.
Time Frame: 0, 180 minutes following administration of the investigational product in crossover phase.
Population: During 2-day cross-over phase, subjects were randomized to receive placebo one day and active on the other. This includes all subjects who received both a placebo and an active dose.
Measure: Mean (Standard Deviation); unit: umol/mL
Groups:
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 5.0g total daily dose of SBI on Day 1 or 5.0g SBI on Day 2 during the double-blind, crossover phase.
  This includes group 1A and 1B.
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 10.0g total daily dose of SBI on Day 1 or 10.0g SBI on Day 2 during the double-blind, crossover phase.
  This includes group 2A and 2B.
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 20.0g total daily dose of SBI on Day 1 or 20.0g SBI on Day 2 during the double-blind, crossover phase.
  This includes group 3A and 3B.
- Placebo: Subjects who will receive a placebo dose(5,10, or 20g) on either day one or two of the crossover phase.
  This includes all subjects who finished the crossover phase, as all subjects received a placebo.
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | Placebo
Number analyzed (Participants) | 18 | 12 | 11 | 41
umol/mL
  Mean - 0 Minutes | 2730.87 (695.33) | 2988.94 (758.92) | 2964.19 (583.50) | 2869.14 (647.01)
  Mean - 180 Minutes: number analyzed (Participants) | 18 | 12 | 11 | 40
  Mean - 180 Minutes | 2723.72 (557.53) | 2785.20 (483.77) | 2893.69 (705.36) | 2736.58 (583.19)

2. Secondary Outcome: Number of Participants With Quantifiable Bovine IgG Plasma Concentration
Description: Plasma samples from participants were tested for bovine IgG content using an ELISA kit with a sheep polyclonal antibody that specifically binds to bovine IgG heavy chain. The limit of quantification was determined to be 3.8 ng/ml and 4.6 ng/ml, in the two separate Elisa kits used (lot numbers 140821 and 140605).
Time Frame: 0 and 90 minutes following investigational product dosing during crossover phase; and after 14 days of open label dosing
Population: Subjects who received at least one dose of SBI. Variations in numbers from the participation flow are due to missing data of certain individuals.
Measure: Count of Participants; unit: Participants
Groups:
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 5.0g total daily dose of SBI on Day 1 or 5.0g SBI on Day 2 during the double-blind crossover phase. Then took 2.5g BID (5.0g daily) during the 14 day open label phase.
  This includes group 1A and 1B.
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 10.0g total daily dose of SBI on Day 1 or 10.0g SBI on Day 2 during the double-blind crossover phase. Then took 5.0g BID (10.0g daily) during the 14 day open label phase.
  This includes group 2A and 2B.
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who will receive either a 20.0g total daily dose of SBI on Day 1 or 20.0g SBI on Day 2 during the double-blind crossover phase. Then took 10.0g BID (20.0g daily) during the 14 day open label phase.
  This includes group 3A and 3B.
- Placebo: Subjects who will receive a placebo dose(5,10, or 20g) on either day one or two of the crossover phase. No open label phase as there is no placebo.
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | Placebo
Number analyzed (Participants) | 18 | 14 | 14 | 42
Participants
  0 minutes: number analyzed (Participants) | 18 | 12 | 11 | 41
  0 minutes | 0 | 0 | 0 | 1
  90 minutes: number analyzed (Participants) | 18 | 12 | 11 | 41
  90 minutes | 0 | 0 | 0 | 1
  Post 14 days of open label dosing: number analyzed (Participants) | 14 | 13 | 12 | 0
  Post 14 days of open label dosing | 0 | 0 | 0 |

3. Secondary Outcome: Bovine IgG Concentration in Stool
Description: Change from baseline in Stool bovine IgG concentration following 14 days of open label dosing.
Time Frame: 14 days after starting the open label phase
Population: Subjects who received at least one dose of product and had at least one stool IgG measurement. No placebo as there is no placebo group in the open label phase.
Measure: Mean (Standard Deviation); unit: pg/mg
Groups:
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who take 2.5g SBI BID (5.0g daily) for 14 days during the open-label phase.
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who take 5.0g SBI BID (10.0g daily) for 14 days during the open-label phase.
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI): Subjects who take 10.0g SBI BID (20.0g daily) for 14 days during the open-label phase.
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI)
Number analyzed (Participants) | 7 | 7 | 7
pg/mg | 100.79 (80.01) | 160.20 (121.09) | 111.59 (76.5)

ADVERSE EVENTS:
Time Frame: 16 Days
Groups:
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase: Subjects that received 5g SBI on either day 1 or day 2 of the crossover phase and reported AE during crossover phase.
  This includes groups 1A and 1B in the crossover phase.
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase: Subjects that received 10g on either day 1 or day 2 of the crossover phase and reported AE during crossover phase.
  This includes groups 2A and 2B in the crossover phase.
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase: Subjects that received 20g on either day 1 or day 2 of the crossover phase and reported AE during crossover phase.
  This includes groups 3A and 3B in the crossover phase.
- Placebo - Crossover Phase: Subjects that received 5, 10, or 20g placebo dose on either day 1 or day 2 of the crossover phase and reported AE during crossover phase. This includes all subjects in the crossover phase.
- 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase: Patients that took 2.5g SBI BID (5g daily) during 14 day open label phase. Reported AE during 14 day open label phase.
  This includes groups 1A and 1B in the open label phase.
- 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase: Patients that took 5g SBI BID (10g daily) during 14 day open label phase. Reported AE during 14 day open label phase.
  This includes groups 2A and 2B in the open label phase.
- 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase: Patients that took 10g SBI BID (20g daily) during 14 day open label phase. Reported AE during 14 day open label phase.
  This includes groups 3A and 3B in the open label phase.
Arm/Group | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase | Placebo - Crossover Phase | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/11 | 0/42 | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/14 | 0/42 | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 4/18 | 0/12 | 3/11 | 0/42 | 7/14 | 4/14 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase (N=18) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase (N=12) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Crossover Phase (N=11) | Placebo - Crossover Phase (N=42) | 5g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase (N=14) | 10g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase (N=14) | 20g Serum-derived Bovine Immunoglobulin Protein Isolate (SBI) - Open Label Phase (N=13)
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — The subject in the 5g-crossover phase section reported the AE at the time they received the placebo dose but 1 day after receiving the SBI dose. This leads to an inconclusive conclusion of what caused this AE.
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in left leg (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flu (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Running nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sore throat (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bloated Feeling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Common Cold (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 — The subject in the 5g-crossover phase section reported the AE at the time they received the placebo dose but 1 day after receiving the SBI dose. This leads to an inconclusive conclusion of what caused this AE.
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 — One subject in the 20g-crossover phase section reported the AE at the time they received the placebo dose but 1 day after receiving the SBI dose. This leads to an inconclusive conclusion of what caused this AE.
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 — The subject in the 5g-crossover phase section reported the AE at the time they received the placebo dose but 1 day after receiving the SBI dose. This leads to an inconclusive conclusion of what caused this AE.
Lightheadedness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gum Shifting (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cramp (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal Cramp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycemia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder Irritation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
45 days